CLINICAL TRIAL: NCT02721381
Title: Comparative Efficacy of a Self-directed and Therapist-assisted Telehealth Parent Training Intervention for Children With ASD
Brief Title: Comparative Efficacy of Self-directed & Therapist-assisted Telehealth Parent Training Intervention for Children With ASD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Brooke Ingersoll, Associate Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R40MC27704
Record Dates: First submitted 2016-03-14; First posted 2016-03-29 (Estimated); Results first posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Parent training; Telehealth; RCT
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Self-Directed Group (Experimental): Participants assigned to the self-directed group will receive access to the secure, password-protected, ImPACT Online web-based program for four months. The web application contains 12, self-directed lessons, each of which takes approximately 75 minutes to complete. Participants will be encouraged to complete one lesson per week and to practice the intervention techniques with their child between each lesson. Each lesson consists of a Narrated Slideshow with embedded video clips, a Written Manual, a self-check quiz, short interactive exercises, a Homework Plan, and reflection questions. Participants in the self-directed group may contact project staff via phone or email for assistance with technology-related problems (e.g., difficulty with logins, problems playing video). However, they will receive no assistance or support in learning the intervention from project staff outside of the self-directed web-based program.
  Interventions: Behavioral: ImPACT Online
- Therapist-Assisted Group (Experimental): Participants assigned to the therapist-assisted group will be given access to the ImPACT Online web-based program for four months and will be encouraged to work through the program at the same pace as the self-directed group. Participants will also receive 2, 30-minute remote coaching sessions per week (24 total sessions) via video conferencing software by a trained therapist to assist them in learning the intervention. The first coaching session of the week will involve the coach and participant and will be used to help clarify the content of the relevant lesson and help the participant apply the lesson content to their own child. The second coaching session of the week will involve the coach, participant, and child and will be used to provide the participant with "live" feedback on their use of the intervention techniques as they practice with their child.
  Interventions: Behavioral: ImPACT Online
- Web-Based Information Control Group (No Intervention): Participants assigned to the web-based information control group will be given access the Resources page with links to the same ASD information websites, but will not receive access to other aspect of the ImPACT Online program. This condition will be used to control for participant maturation as well as the potentially confounding effect of having access to autism-related information via the internet.

INTERVENTIONS:
Behavioral: ImPACT Online — ImPACT Online is an interactive, web-based telehealth intervention that teaches parents to promote their child's social-communication skills during play and daily routines. The intervention content was adapted from Project ImPACT, a manualized parent training curriculum that uses a blend of developmental and naturalistic behavioral intervention techniques, including following the child's lead, imitating the child, using heightened animation, using simplified language around the child's focus of attention, environmental arrangement strategies, prompting, and natural reinforcement during child-directed activities. There is strong empirical support for the intervention techniques for increasing social communication in children, increasing parent fidelity, and child language skills.
  Arms: Self-Directed Group; Therapist-Assisted Group

SUMMARY:
The specific objectives of this project are to conduct a randomized control trial to examine the effect of a novel, telehealth parent training intervention for children with autism spectrum disorder (ASD), ImPACT Online, on parent and child outcomes. The investigators will compare the benefits of the self-directed and therapist-assisted delivery formats, and examine moderators and mediators of treatment outcomes. The investigators anticipate that both the self-directed and therapist-assisted models of ImPACT Online will be effective methods for teaching parents to use evidence-based intervention strategies and for increasing parent self-efficacy compared to a web-based information control group. Participants will be randomly assigned to one of three groups. One-third of participants will be in the therapist-assisted group; one-third will be in the self-directed group; and one-third will be in a web-based information control group.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a chronic and pervasive neurodevelopmental disorder characterized by deficits in social communication and the presence of restricted and repetitive behaviors. Individuals with ASD often require intensive and comprehensive intervention across the life span. There has been a dramatic increase in the number of individuals with this diagnosis over the last two decades, with current prevalence rates as high as 1 in 68. However, there has not been corresponding growth in the availability of evidence-based intervention services, contributing to high levels of unmet service needs for individuals with ASD and their families. The vast majority of families of children with ASD report receiving substantially fewer hours of services than recommended by the National Research Council. Furthermore, levels of unmet service needs are even higher for families residing in rural and medically underserved communities. Thus, systematic research focused on developing and improving strategies for dissemination and implementation of evidence-based ASD services is a high priority, particularly for chronically underserved communities.

Parent training programs are one cost-effective and ecologically valid way to increase access to evidence-based ASD intervention. Training parents to provide intervention themselves can increase the number of intervention hours a child receives and improve child outcomes. A number of studies have demonstrated that parents can learn to use evidence-based intervention strategies with a high degree of fidelity and their children experience gains in language and social communication development, decreases in disruptive behavior, and greater generalization and maintenance of child skill. These benefits are recognized by parents, who report parent training to be the most effective practice for promoting their child's overall development. Parent training also improves family quality of life by increasing parent self-efficacy and reducing parenting stress, which is particularly important given the high rate of stress and depression found in parents of children with ASD.

Despite these benefits, there continue to be barriers to the dissemination of training to parents. Formal parent training programs are rare in community-based early intervention settings for young children with ASD. For example, in a recent North Carolina survey, only 8% of parents of children with ASD under 4 reported receiving parent training. Barriers to the provision of parent training include a shortage of trained professionals, lengthy waitlists, limited financial resources and transportation, lack of child care, geographic isolation, and time limitations. These barriers may be even more pronounced for families who live in rural areas, for whom long distances, poor roads, and climatic barriers limit the ability of parents to receive services. Thus, it is essential to consider the adaptation of evidence-based parent training programs to non-traditional service delivery models to increase access to services.

Telehealth, or the provision of health services and information through the Internet and related technologies, has the potential to replace or, at the very least, augment traditional service models to increase access to evidence-based services. Users of telehealth programs are able to interact directly with instructional content through video, animation, and active learning tasks, as well as with other individuals, including expert clinicians, via email and teleconferencing systems. The number of individuals with access to internet-based technologies has grown considerably in recent years (File T, 2013), and it is now estimated that 75% of U.S. households have a home computer with high-speed internet, and nearly 87% of adults are able to access the internet from home, work, or elsewhere. Telehealth services are becoming increasingly common with over 3,000 U.S. sites using distance-based service delivery models to provide patient care.

Telehealth programs can reduce patient and provider costs and increase provider system coverage relative to traditional in-person service delivery models. Such programs have been shown to greatly improve care for patients with chronic diseases, such as diabetes, heart disease, and asthma, and increase access to evidence-based health promotion (i.e., smoking cessation, dietary change, physical activity), psychological (i.e., CBT for depression and anxiety), and parenting interventions. Patients are often very satisfied with the care they receive through telehealth services, and efficacy studies have found moderate to large effects of telehealth interventions on participant knowledge and behavior change. Further, several recent meta-analyses have found that CBT delivered via telehealth is as effective as traditional therapist-delivered intervention. Taken together, these data suggest that telehealth may serve as a promising alternative service delivery model to increase the dissemination of ASD parent training programs.

Telehealth interventions can be either self-directed, in which the participant engages with the interactive program at his or her own pace, or therapist-assisted, in which the participant receives additional guidance from a trained professional as he or she completes the program. Self-directed programs have far greater dissemination potential as they do not require a trained professional and can typically be administered at a much reduced cost. At the same time, research on telehealth CBT interventions for mood and anxiety have found that therapist-assisted programs lead to better client outcomes than self-directed programs. This finding may be particularly relevant for telehealth parent training interventions, as research suggests that parent coaching is important for increasing parents' fidelity of implementation, and coaching is a core component of existing evidence-based parent training interventions for children with ASD.

There has been growing interest in extending telehealth interventions to parent training for children with ASD; yet empirical evaluations of such programs are very limited. Several uncontrolled studies of self-directed telehealth parent training programs have shown that parents of children with ASD find such programs to be highly acceptable, and program use is associated with gains in parent knowledge of evidence-based intervention procedures. Preliminary empirical studies have suggested that parents can learn to implement evidence-based intervention techniques with fidelity after using a self-directed telehealth parent training program. A small controlled study found that parents who were given access to a DVD-based self-directed program made greater gains in their correct use of pivotal response training (PRT) strategies, provided their children with more language opportunities, and displayed greater confidence in parent-child interactions, than parents in a no-treatment control group. Using a single-subject design, demonstrated that parents improved their correct use of reciprocal imitation training (RIT) techniques after completing a web-based, self-directed program. However, one third of the participants required additional in-person coaching in order to meet the pre-determined fidelity of implementation criterion. In both studies, improvements in child behaviors targeted by the interventions were also observed. Importantly, parents in both studies indicated that immediate feedback or coaching from an expert clinician would have been a helpful addition to the program.

Several recent single-subject design studies have examined the efficacy of therapist-assisted telehealth parent training programs for children with ASD. Researchers examined the effect of both a DVD-based and web-based program in conjunction with weekly remote coaching sessions via video-conferencing to teach parents the Early Start Denver Model (ESDM). Results suggested that parents increased their correct usage of the intervention strategies and altered their engagement styles to be more attentive and responsive to their children after the therapist-assisted telehealth program. Furthermore, children in both studies demonstrated gains in important social communicative behaviors (e.g., language, imitative behaviors). In an attempt to evaluate the relative contributions of self-directed instruction and remote coaching on parent learning of RIT, researchers conducted a second study that measured parents' use of RIT techniques with their child prior to completing a self-directed, web-based program, after completing the self-directed program but before receiving remote coaching via video-conferencing, and after receiving remote coaching. Similar to their previous study, all parents improved their correct use of the intervention techniques in response to the self-directed program, but roughly a third showed additional benefit from the provision of remote coaching. In addition, most children demonstrated gains in imitation skills (the target of the intervention) with the onset of treatment; however, child gains were most robust during the coaching portion of the program.

These preliminary findings suggest telehealth parent training interventions are highly acceptable to parents of children with ASD, and can result in improvements in parent knowledge and implementation of evidence-based intervention techniques and gains in child social communication skills. To date, no studies have conducted a head-to-head comparison of self-directed and therapist-assisted telehealth parent training interventions. However, data thus far indicate that parent coaching may be necessary for some, but not all parents to successfully implement evidence-based intervention techniques with fidelity. A more nuanced appreciation of the contributions offered by each component, as well as which parents are more likely to benefit from each, will make it possible to develop more cost-effective delivery models in which services can be offered at different levels of intensity, depending on specific needs of the family (i.e., stepped-care).

ImPACT Online is an interactive, web-based telehealth intervention that teaches parents to promote their child's social-communication skills during play and daily routines. The intervention content was adapted from Project ImPACT, a manualized parent training curriculum that uses a blend of developmental and naturalistic behavioral intervention techniques, including following the child's lead, imitating the child, using heightened animation, using simplified language around the child's focus of attention, environmental arrangement strategies, prompting, and natural reinforcement during child-directed activities. There is strong empirical support for the intervention techniques for increasing social communication in children with ASD. In addition, several studies have demonstrated the efficacy of the original parent training curriculum for increasing parent fidelity and child language skills.

The original curriculum was designed to be implemented over 12 weeks in either an individual or group format by an in-person parent trainer. The investigators have adapted the program so that the intervention content is presented in 12 interactive, web-based modules or lessons. These lessons can be administered as a standalone intervention (self-directed model) or in combination with remote coaching (therapist-assisted model). Program development was guided by the technology acceptance model56, media richness theory57,58, and principles of instructional design59. To ensure usability, The investigators used an iterative development process with input from focus groups of parents and intervention providers, and interviews with pilot participants. The investigators have conducted a feasibility trial of the self-directed and therapist-assisted models with 25 families, the majority of whom (75%) reside in rural and medically underserved areas. Our data thus far strongly support the acceptability and feasibility of the web-based modules and the remote coaching protocol, and suggest that such models can be used to effectively reach individuals residing in underserved communities. Further, our data lend preliminary support for the positive effect of the program on parent fidelity of implementation, self-efficacy, and child language. The next step in evaluating ImPACT Online is to conduct a fully-powered RCT with a control group to evaluate the comparative efficacy of the self-directed and therapist-assisted telehealth intervention models on key parent and child behaviors, as well as to examine potential mediators and moderators of treatment outcomes.

Statement of the Problem Research indicates that early, intensive intervention can lead to significant improvements for children with ASD. There has been a dramatic increase in the prevalence of ASD over the past two decades, but not a corresponding growth in availability of evidence-based intervention services. This has led to high levels of unmet service needs for individuals with ASD and their families. Parent training is one cost-effective and ecologically valid approach to increase access to intervention. Additional benefits include increases in parenting self-efficacy and decreases in parenting stress. Yet, there continue to be barriers involved with the dissemination of training to parents. Telehealth interventions have the potential to replace, or at the least augment, traditional service models to increase access to evidence-based services, particularly in rural and medically underserved areas. There is increasing evidence to suggest that such programs can reduce patient and provider costs and increase provider system coverage relative to traditional in-person service delivery models.

Although there has been growing interest in extending telehealth interventions to parent training for children with ASD, empirical evaluations of such programs are limited, and little is known regarding the relative benefits of self-directed and therapist-assisted telehealth interventions for ASD. Self-directed programs have far greater dissemination potential as they do not require a trained professional and can typically be administered at a much reduced cost. At the same time, research on telehealth interventions for other disorders have found that therapist-assisted programs lead to better client outcomes than self-directed programs. A better understanding of the relative benefits of these two delivery formats on parent and child outcomes, as well as the families for whom each format is most and least effective, is crucial for the development of effective and efficient telehealth parent training interventions.

The specific objectives of this project are to conduct a randomized control trial to examine the effect of a novel, telehealth parent training intervention for children with autism spectrum disorder (ASD), ImPACT Online, on parent and child outcomes. The investigators will compare the benefits of the self-directed and therapist-assisted delivery formats, and examine moderators and mediators of treatment outcomes. The investigators anticipate that both the self-directed and therapist-assisted models of ImPACT Online will be effective methods for teaching parents to use evidence-based intervention strategies and for increasing parent self-efficacy compared to a web-based information control group. Parents' use of these strategies will greatly enhance the amount of evidence-based intervention that their children receive and improve generalization and maintenance of skills, positively impacting their children's language development. The investigators anticipate that parents in the therapist-assisted group will outperform parents in the self-directed group on the primary parent outcome measures at the group level; however, our moderator analyses may indicate parents for whom each approach is more and less effective. These data will be key to informing a stepped-care model in which parents can be offered the intervention at different levels of intensity (self-directed or therapist-assisted), depending on the specific needs of the family. Further, if this approach to parent training is successful, it has the potential to greatly increase access to evidence-based intervention for children with ASD, especially those living in rural and underserved areas.

Ninety families of young children with ASD will be assessed at pre-treatment (T1), randomized to the self-directed ImPACT Online, therapist-assisted ImPACT Online, or web-based information control condition, and will receive treatment for 4 months. Outcome assessments will occur at post-treatment (T2) and a 3-month follow-up (T3).

Aim 1: To examine the comparative efficacy of self-directed and therapist-assisted ImPACT Online on parent outcomes at post-treatment and the 3-month follow-up. The primary goal of ImPACT Online is to teach parents to use specific intervention techniques to promote their child's social communication development. As parents gain the knowledge and skills to help their child, their self-efficacy as a parent is expected to increase. Thus, The investigators will compare the effects of the two telehealth intervention models on parent fidelity and parent self-efficacy at post-treatment and a 3-month follow-up. It is hypothesized that families randomized to either of the two telehealth conditions will demonstrate greater gains in parent fidelity and parent self-efficacy at post-treatment and 3-month follow-up than parents assigned to the control group. Given research on telehealth interventions for other disorders suggesting an added benefit of therapist-assistance, it is hypothesized that families randomized to the therapist-assisted telehealth condition will demonstrate greater gains in parent outcomes relative to parents in the self-directed telehealth condition at post and follow-up.

Aim 2: To examine the comparative efficacy of self-directed and therapist-assisted ImPACT Online on child outcomes at the 3-month follow-up. Parent use of the intervention techniques over time is expected to lead to improvements in child verbal language. Thus, The investigators will compare the effects of the two intervention models on child verbal language at the 3-month follow-up. It is hypothesized that families randomized to either of the two telehealth conditions will demonstrate greater gains in child verbal language at follow-up than parents assigned to the control group. Given the stronger effects on parent outcomes expected for the therapist-assisted intervention, it is hypothesized that families randomized to the therapist-assisted telehealth condition will demonstrate greater gains in child verbal language relative to parents in the self-directed telehealth condition at follow-up.

Aim 3: To examine whether pre-treatment parenting stress moderates the effects of ImPACT Online on parent fidelity and parent self-efficacy at post-treatment. Our goal is to identify the families for whom the different telehealth delivery formats are most and least effective. Prior research has indicated a negative association between pre-treatment parenting stress levels and treatment outcomes in ASD parent training interventions. Thus, The investigators will examine pre-treatment parenting stress as a putative moderator of parent treatment response. It is hypothesized that the effects of ImPACT Online on parent fidelity and parent self-efficacy will be stronger for parents with lower pre-treatment levels of parenting stress. It is anticipated that pre-treatment parenting stress levels may also differentially impact parent outcomes for the two telehealth delivery formats. For example, high levels of pre-treatment parenting stress may be more likely to negatively impact parent outcomes in the self-directed group, because parents do not have the additional support of a coach. Thus, it is also hypothesized that the relationship between parenting stress and parent outcomes will be stronger in the self-directed group than the therapist-assisted group.

Aim 4: To examine whether gains in parent fidelity and parent self-efficacy at post-treatment mediate the effects of the ImPACT Online on child verbal language at the 3-month follow-up. In ASD parent training studies it has been assumed that improvements in child outcomes are a result of improvements in their parents' ability to implement the treatment. However, this relationship has rarely been directly tested. While parent fidelity is a likely candidate, it is also possible that changes in other important parent behaviors, such as parent self-efficacy, may be important factors in promoting child change. For example, it may be that parents who feel more self-efficacious in the parenting role may engage with their child more often, have higher expectations for their child's behavior, or may more effectively advocate for their child's needs, all of which might result in "non-specific" treatment effects. Thus, The investigators will examine mediators of child changes to better understand how our parent training model is affecting child outcomes. Specifically, The investigators will examine whether improvements in child verbal language as a result of treatment are mediated by changes in parent fidelity and/or parent self-efficacy. It is hypothesized that the effects of ImPACT Online on child verbal language at the 3-month follow-up will be greater for children whose parents demonstrate greater gains in parent fidelity and parent self-efficacy from pre- to post-treatment.

Aim 5 (exploratory): To identify predictors of adherence to ImPACT Online. In order to fully capitalize on the benefits of telehealth, it is important to understand factors that influence parent adherence to ImPACT Online. The investigators have selected one program-level (therapist assistance) and three individual-level (computer/internet fluency, parent expectancies, treatment acceptability) factors that have been found to influence adherence to parent training and/or telehealth-based interventions in previous work. The investigators will also examine whether any sociodemographic variables predict treatment adherence. It is hypothesized that therapist assistance will predict adherence, such the therapist-assisted group will exhibit greater adherence than the self-directed group, and that computer/internet fluency, parent expectancy, and treatment acceptability will be positively associated with adherence to ImPACT online. Finally, The investigators hypothesize that some sociodemographic variable will be found to predict treatment adherence.

Research Design and Methods Participants. 90 children with ASD between the ages of 18 and 72 months will be recruited for this study. This sample size was determined to be adequate for maintaining adequate power for the proposed statistical analyses, while allowing for some attrition. To ensure that the sample includes a sufficient number of participants who are traditionally underserved, The investigators will oversample for participants living in a federally designated rural and/or medically-underserved area, and those with additional risk factors associated with decreased access to care, including low parental education, single-parent household, racial or ethnic minority, and immigrant status. To be eligible, children must receive a DSM-V-informed clinical diagnosis of Autism Spectrum Disorder based on the Autism Diagnostic Observation Schedule (ADOS). In light of research suggesting that diagnostic stability is lower in children under 30 months. Results of diagnostic testing for the younger children in our sample will be interpreted cautiously and discussed with parents in a sensitive and transparent manner. Children with a history of significant brain injury, known neurological or genetic condition, significant sensory or motor impairment, or major medical problems will be excluded as they might be expected to respond differently than children with ASD only or require program modifications.

Participants will be recruited through our ongoing contacts with community agencies and professionals serving young children with ASD in Michigan. The P.I. has extensive experience recruiting families of young children with ASD for intervention studies. Previous research efforts, including a pilot RCT of ImPACT Online, strongly suggest that The investigators will be able to recruit the proposed number of participants. The MSU Autism Lab uses a number of strategies to ensure retention, including maintaining responsive relationships with participating families, providing clinical consultation and referral, and maintaining contact through newsletters and periodic family outings. Retention rates for previous studies, including the pilot RCT of this intervention, have all been above 90%.

Group assignment. It is possible that group differences in child age and/or developmental quotient (DQ) at intake could affect the internal validity of the study. Thus, participants will be stratified by age (18-35 months; 36-72 months) and developmental quotient (DQ<50; DQ≥50) prior to being randomized. After stratification by age and DQ, participants will be randomly assigned to the one of the three groups using random permuted blocks of 6. This approach has been shown to yield groups that are closely balanced with regard to size and relevant pre-treatment characteristics. All pre-treatment assessments will be collected prior to randomization to prevent bias during testing based on knowledge of future group placement.

Children in all three groups will continue to receive their existing educational programming. It is not expected that non-treatment intervention participation will differ systematically across groups; however, information on the amount and type of outside services and changes to services will be collected for each child on a monthly basis throughout their participation. All families who express a need for a computer or high speed internet will be provided with a loaner laptop and a high speed internet service plan for the duration of their participation.

Training plan and coaching fidelity for Therapist-Assisted Group. Therapists who provide the remote coaching will be masters' level project staff trained to fidelity in the coaching procedure by the PI. Training includes a combination of didactic training, observation of remote coaching sessions, role play, and hands-on coaching during practice with children with ASD and their parents. All therapists will be required to establish fidelity with non-study participants prior to beginning the study, as determined by >90% correct implementation on the Coaching Fidelity Checklist (Ingersoll & Dvortcsak, 2010). This training approach has been highly successful for ensuring fidelity of therapists. Coaching fidelity data will be collected for a randomly selected sample of 20% of sessions and analyzed to ensure correct implementation of the remote coaching procedure. If a therapist falls below 90% correct implementation, the PI will provide additional training and feedback until the therapist re-establishes fidelity.

Assessment protocol. Participants in each group will receive assessments at 3 time points: pre-treatment (prior to randomization) (T1), post-treatment (T2), and 3-month follow-up (T3). A 3-month follow-up was chosen to allow time for the children to beneﬁt from their parents' use of the intervention strategies, while ensuring that follow-up assessments for all children can be completed within the project period. Each assessment period will consist of three to four hours of testing, involving direct child assessment, home observation of a parent-child interaction, and parent-report measures of parent and child functioning which will be completed in the family home.

Examiners who are blind to the study objectives and treatment group assignment will conduct all assessments. Assessments requiring behavioral coding will be videotaped and scored by trained observers who are blind to treatment condition. One-third of the assessments will be coded by a second, independent observer to determine interobserver agreement. Families will be compensated $25 per assessment period ($75 per family).

ELIGIBILITY:
Inclusion Criteria for child participants:

* a DSM-V-informed clinical diagnosis of Autism Spectrum Disorder based on the Autism Diagnostic Observation Schedule (ADOS)

Exclusion Criteria for child participants:

* history of significant brain injury, known neurological or genetic condition
* significant sensory or motor impairment
* major medical problems

Inclusion Criteria for parent participants:

* primary caregiver of child participant
* Proficient in English

Exclusion Criteria for parent participants:

-under 18 years

Ages: 18 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brooke Ingersoll, PhD, Principal Investigator — Michigan State University
Locations (1):
- Michigan State University Autism Lab, East Lansing, Michigan, United States

REFERENCES:
- [Background] American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders. 5th ed. Arlington, VA: American Psychiatric Publishing; 2013.
- [Background] National Research Council. Educating Children With Autism. Washington, DC: National Academy Press; 2001.
- [Background] Developmental Disabilities Monitoring Network Surveillance Year 2010 Principal Investigators; Centers for Disease Control and Prevention (CDC). Prevalence of autism spectrum disorder among children aged 8 years - autism and developmental disabilities monitoring network, 11 sites, United States, 2010. MMWR Surveill Summ. 2014 Mar 28;63(2):1-21. PMID 24670961
- [Background] Bitterman A, Daley TC, Misra S, Carlson E, Markowitz J. A national sample of preschoolers with autism spectrum disorders: special education services and parent satisfaction. J Autism Dev Disord. 2008 Sep;38(8):1509-17. doi: 10.1007/s10803-007-0531-9. Epub 2008 Jan 29. PMID 18228122
- [Background] Kogan MD, Strickland BB, Blumberg SJ, Singh GK, Perrin JM, van Dyck PC. A national profile of the health care experiences and family impact of autism spectrum disorder among children in the United States, 2005-2006. Pediatrics. 2008 Dec;122(6):e1149-58. doi: 10.1542/peds.2008-1057. PMID 19047216
- [Background] Hume K, Bellini S, Pratt C. The usage and perceived outcomes of early intervention and early childhood programs for young children with Autism Spectrum Disorder. Topics Early Child Spec Educ. 2005;25(4):195-207.
- [Background] Thomas KC, Ellis AR, McLaurin C, Daniels J, Morrissey JP. Access to care for autism-related services. J Autism Dev Disord. 2007 Nov;37(10):1902-12. doi: 10.1007/s10803-006-0323-7. Epub 2007 Mar 19. PMID 17372817
- [Background] Mandell DS, Novak MM, Zubritsky CD. Factors associated with age of diagnosis among children with autism spectrum disorders. Pediatrics. 2005 Dec;116(6):1480-6. doi: 10.1542/peds.2005-0185. PMID 16322174
- [Background] Ingersoll BR, Wainer AL. Pilot study of a school-based parent training program for preschoolers with ASD. Autism. 2013 Jul;17(4):434-48. doi: 10.1177/1362361311427155. Epub 2011 Nov 15. PMID 22087044
- [Background] Kaiser AP, Hancock TB, Nietfeld JP. Early education and development: The effects of parent-implemented Enhanced Milieu Teaching on the social communication of children who have Autism. Early Educ Dev. 2010;11(4):423-446. doi:10.1207/s15566935eed1104.
- [Background] Vismara LA, Colombi C, Rogers SJ. Can one hour per week of therapy lead to lasting changes in young children with autism? Autism. 2009 Jan;13(1):93-115. doi: 10.1177/1362361307098516. PMID 19176579
- [Background] Bearss K, Johnson C, Handen B, Smith T, Scahill L. A pilot study of parent training in young children with autism spectrum disorders and disruptive behavior. J Autism Dev Disord. 2013 Apr;43(4):829-40. doi: 10.1007/s10803-012-1624-7. PMID 22941342
- [Background] Moes DR, Frea WD. Contextualized behavioral support in early intervention for children with autism and their families. J Autism Dev Disord. 2002 Dec;32(6):519-33. doi: 10.1023/a:1021298729297. PMID 12553589
- [Background] Koegel RL, Bimbela A, Schreibman L. Collateral effects of parent training on family interactions. J Autism Dev Disord. 1996 Jun;26(3):347-59. doi: 10.1007/BF02172479. PMID 8792265
- [Background] Sofronoff K, Farbotko M. The effectiveness of parent management training to increase self-efficacy in parents of children with Asperger syndrome. Autism. 2002 Sep;6(3):271-86. doi: 10.1177/1362361302006003005. PMID 12212918
- [Background] Tonge B, Brereton A, Kiomall M, Mackinnon A, King N, Rinehart N. Effects on parental mental health of an education and skills training program for parents of young children with autism: a randomized controlled trial. J Am Acad Child Adolesc Psychiatry. 2006 May;45(5):561-569. doi: 10.1097/01.chi.0000205701.48324.26. PMID 16670650
- [Background] Estes A, Munson J, Dawson G, Koehler E, Zhou XH, Abbott R. Parenting stress and psychological functioning among mothers of preschool children with autism and developmental delay. Autism. 2009 Jul;13(4):375-87. doi: 10.1177/1362361309105658. PMID 19535467
- [Background] Thomas KC, Morrissey JP, McLaurin C. Use of autism-related services by families and children. J Autism Dev Disord. 2007 May;37(5):818-29. doi: 10.1007/s10803-006-0208-9. PMID 17146709
- [Background] Stahmer AC, Gist K. The effects of an accelerated parent education program on technique mastery and child outcome. J Posit Behav Interv. 2001;3(2):75-82. doi:10.1177/109830070100300203.
- [Background] Symon JB. Expanding interventions for children with Autism: Parents as trainers. J Posit Behav Interv. 2005;7(3):159-173. doi:10.1177/10983007050070030501.
- [Background] Connell S, Sanders MR, Markie-Dadds C. Self-directed behavioral family intervention for parents of oppositional children in rural and remote areas. Behav Modif. 1997 Oct;21(4):379-408. doi: 10.1177/01454455970214001. PMID 9337598
- [Background] Baggett KM, Davis B, Feil EG, Sheeber LB, Landry SH, Carta JJ, Leve C. Technologies for expanding the reach of evidence-based interventions: Preliminary results for promoting social-emotional development in early childhood. Topics Early Child Spec Educ. 2010 Feb 1;29(4):226-238. doi: 10.1177/0271121409354782. No abstract available. PMID 20454545
- [Background] United States Department of Education, Office of Planning, Evaluation, and Policy Development. Evaluation of Evidence-Based Practices in Online Learning: A Meta-Analysis and Review of Online Learning Studies. Washington, DC; 2010.
- [Background] Weingardt KR. The role of instructional design and technology in the dissemination of empirically supported, manual-based therapies. Clin Psychol Scienec Pract. 2004;11:2004.
- [Background] File T. Computer and internet use in the United States: Population characteristics. Washington, DC: US Census Bureau; 2013.
- [Background] Bureau USC. Statistical abstract of the United States: 2013. 2013.
- [Background] Internet User Demographics. Pew Res Cent Internet Proj Surv January 9-12, 2014. 2014.
- [Background] Association AT. What is telemedicine? 2013.
- [Background] Gros DF, Morland LA, Greene CJ, et al. Delivery of evidence-based psychotherapy via video telehealth. J Psychopathol Behav Assess. 2013;35(4):506-521. doi:10.1007/s10862-013-9363-4.
- [Background] Wootton R. Twenty years of telemedicine in chronic disease management--an evidence synthesis. J Telemed Telecare. 2012 Jun;18(4):211-20. doi: 10.1258/jtt.2012.120219. PMID 22674020
- [Background] Krebs P, Prochaska JO, Rossi JS. A meta-analysis of computer-tailored interventions for health behavior change. Prev Med. 2010 Sep-Oct;51(3-4):214-21. doi: 10.1016/j.ypmed.2010.06.004. Epub 2010 Jun 15. PMID 20558196
- [Background] Andersson G, Cuijpers P. Internet-based and other computerized psychological treatments for adult depression: a meta-analysis. Cogn Behav Ther. 2009;38(4):196-205. doi: 10.1080/16506070903318960. PMID 20183695
- [Background] Nieuwboer CC, Fukkink RG, Hermanns JMA. Online programs as tools to improve parenting: A meta-analytic review. Child Youth Serv Rev. 2013;35(11):1823-1829. doi:10.1016/j.childyouth.2013.08.008.
- [Background] Gustke SS, Balch DC, West VL, Rogers LO. Patient satisfaction with telemedicine. Telemed Journal2. 2000;6(1):5-13.
- [Background] Mair F, Whitten P. Systematic review of studies of patient satisfaction with telemedicine. BMJ. 2000 Jun 3;320(7248):1517-20. doi: 10.1136/bmj.320.7248.1517. PMID 10834899
- [Background] Andrews G, Cuijpers P, Craske MG, McEvoy P, Titov N. Computer therapy for the anxiety and depressive disorders is effective, acceptable and practical health care: a meta-analysis. PLoS One. 2010 Oct 13;5(10):e13196. doi: 10.1371/journal.pone.0013196. PMID 20967242
- [Background] Reger MA, Gahm GA. A meta-analysis of the effects of internet- and computer-based cognitive-behavioral treatments for anxiety. J Clin Psychol. 2009 Jan;65(1):53-75. doi: 10.1002/jclp.20536. PMID 19051274
- [Background] Spek V, Cuijpers P, Nyklicek I, Riper H, Keyzer J, Pop V. Internet-based cognitive behaviour therapy for symptoms of depression and anxiety: a meta-analysis. Psychol Med. 2007 Mar;37(3):319-28. doi: 10.1017/S0033291706008944. Epub 2006 Nov 20. PMID 17112400
- [Background] Kaminski JW, Valle LA, Filene JH, Boyle CL. A meta-analytic review of components associated with parent training program effectiveness. J Abnorm Child Psychol. 2008 May;36(4):567-89. doi: 10.1007/s10802-007-9201-9. Epub 2008 Jan 19. PMID 18205039
- [Background] Kaiser AP, Hemmeter ML, Ostrosky MM, Alpert CL, Hancock TB. The effects of group training and individual feedback on parent use of Milieu Teaching. Commun Disord Q. 1995;16(2):39-48. doi:10.1177/152574019501600206.
- [Background] Steiner AM, Koegel LK, Koegel RL, Ence WA. Issues and theoretical constructs regarding parent education for autism spectrum disorders. J Autism Dev Disord. 2012 Jun;42(6):1218-27. doi: 10.1007/s10803-011-1194-0. PMID 21336525
- [Background] Hamad CD, Serna RW, Morrison L, Fleming R. Extending the Reach of Early Intervention Training for Practitioners: A Preliminary Investigation of an Online Curriculum for Teaching Behavioral Intervention Knowledge in Autism to Families and Service Providers. Infants Young Child. 2010 Jul 1;23(3):195-208. doi: 10.1097/IYC.0b013e3181e32d5e. PMID 23504540
- [Background] Howroyd C, Peeters T. Parent participation in early intervention with software-assited guidance from AutismPro. Good Autism Pract. 2007;8(2):31-36.
- [Background] Kobak KA, Stone WL, Wallace E, Warren Z, Swanson A, Robson K. A web-based tutorial for parents of young children with autism: results from a pilot study. Telemed J E Health. 2011 Dec;17(10):804-8. doi: 10.1089/tmj.2011.0060. Epub 2011 Oct 19. PMID 22011005
- [Background] Jang J, Dixon DR, Tarbox J, Granpeesheh D, Kornack J, de Nocker Y. Randomized trial of an eLearning program for training family members of children with autism in the principles and procedures of applied behavior analysis. Res Autism Spectr Disord. 2012;6(2):852-856. doi:10.1016/j.rasd.2011.11.004.
- [Background] Nefdt N, Koegel R, Singer G, Gerber M. The use of a self-directed learning program to provide introductory training in Pivotal Response Treatment to parents of children with Autism. J Posit Behav Interv. 2009;12(1):23-32. doi:10.1177/1098300709334796.
- [Background] Wainer AL, Ingersoll BR. Disseminating ASD interventions: a pilot study of a distance learning program for parents and professionals. J Autism Dev Disord. 2013 Jan;43(1):11-24. doi: 10.1007/s10803-012-1538-4. PMID 22547028
- [Derived] Ingersoll B, Frost KM, Straiton D, Ramos AP, Casagrande K. Telehealth coaching in Project ImPACT indirectly affects children's expressive language ability through parent intervention strategy use and child intentional communication: An RCT. Autism Res. 2024 Oct;17(10):2177-2187. doi: 10.1002/aur.3230. Epub 2024 Sep 4. PMID 39233512

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place in Michigan and focused on underserved communities as defined by residence in a Rural Health and/or Health Provider Shortage Area by the U.S. Health Resource & Services Administration; however, families did not have to live in an underserved community to be enrolled.
Groups:
- Parent: Self-Directed Group: Parent participants assigned to the self-directed group will receive access to the secure, password-protected, ImPACT Online web-based program for four months. The intervention content was adapted from Project ImPACT, a manualized NDBI parent training curriculum. The web application contains 12, self-directed lessons, each of which takes approximately 75 minutes to complete. Parent participants will be encouraged to complete one lesson per week and to practice the intervention techniques with their child between each lesson. Each lesson consists of a Narrated Slideshow with embedded video clips, a Written Manual, a self-check quiz, short interactive exercises, a Homework Plan, and reflection questions. Parent participants in the self-directed group may contact project staff via phone or email for assistance with technology-related problems (e.g., difficulty with logins, problems playing video). However, they will receive no assistance or support in learning the intervention from project staff outside of the self-directed web-based program.
- Child: Self-Directed Group: Child participants will receive Project ImPACT intervention from their parent as trained in the self-directed group.
- Parent: Therapist-Assisted Group: Parent participants assigned to the therapist-assisted group will be given access to the ImPACT Online web-based program for four months and will be encouraged to work through the program at the same pace as the self-directed group. The intervention content was adapted from Project ImPACT, a manualized NDBI parent training curriculum. Parent participants will also receive 2, 30-minute remote coaching sessions per week (24 total sessions) via video conferencing software by a trained therapist to assist them in learning the intervention. The first coaching session of the week will involve the coach and participant and will be used to help clarify the content of the relevant lesson and help the parent participant apply the lesson content to their own child. The second coaching session of the week will involve the coach, participant, and child and will be used to provide the participant with "live" feedback on their use of the intervention techniques as they practice with their child.
- Child: Therapist-Assisted Group: Child participants will receive Project ImPACT intervention from their parent as trained in the therapist-assisted group.
- Parent: Information and Resource Support Control Group: Parent participants assigned to the web-based information control group will be given access the Resources page with links to the same ASD information websites, but will not receive access to other aspect of the ImPACT Online program. This condition will be used to control for child participant maturation as well as the potentially confounding effect of parent participants having access to autism-related information via the internet.
- Child: Information and Resource Support Group: Child participants will interact with their parent without training in Project ImPACT.
Period: Overall Study
Arm/Group | Parent: Self-Directed Group | Child: Self-Directed Group | Parent: Therapist-Assisted Group | Child: Therapist-Assisted Group | Parent: Information and Resource Support Control Group | Child: Information and Resource Support Group
Started | 24 | 24 | 22 | 22 | 19 | 19
Completed | 21 | 21 | 21 | 21 | 17 | 17
Not Completed | 3 | 3 | 1 | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Parent: Self-Directed Group: Parent participants assigned to the self-directed group will receive access to the secure, password-protected, ImPACT Online web-based program for four months. The intervention content was adapted from Project ImPACT, a manualized NDBI parent training curriculum. The web application contains 12, self-directed lessons, each of which takes approximately 75 minutes to complete. Parent participants will be encouraged to complete one lesson per week and to practice the intervention techniques with their child between each lesson. Each lesson consists of a Narrated Slideshow with embedded video clips, a Written Manual, a self-check quiz, short interactive exercises, a Homework Plan, and reflection questions. Participants in the self-directed group may contact project staff via phone or email for assistance with technology-related problems (e.g., difficulty with logins, problems playing video). However, they will receive no assistance or support in learning the intervention from project staff outside of the self-directed web-based program.
- Parent: Therapist-Assisted Group: Parent participants assigned to the therapist-assisted group will be given access to the ImPACT Online web-based program for four months and will be encouraged to work through the program at the same pace as the self-directed group. The intervention content was adapted from Project ImPACT, a manualized NDBI parent training curriculum. Parent participants will also receive 2, 30-minute remote coaching sessions per week (24 total sessions) via video conferencing software by a trained therapist to assist them in learning the intervention. The first coaching session of the week will involve the coach and participant and will be used to help clarify the content of the relevant lesson and help the parent participant apply the lesson content to their own child. The second coaching session of the week will involve the coach, parent participant, and child participant and will be used to provide the participant with "live" feedback on their use of the intervention techniques as they practice with their child.
- Child: Information and Resource Support: Child participants will interact with their parent without training in Project ImPACT.
- Total: Total of all reporting groups
Arm/Group | Parent: Self-Directed Group | Child: Self-Directed Group | Parent: Therapist-Assisted Group | Child: Therapist-Assisted Group | Parent: Information and Resource Support Control Group | Child: Information and Resource Support | Total
Number analyzed (Participants) | 24 | 24 | 22 | 22 | 19 | 19 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 24 | 0 | 22 | 0 | 19 | 65
  Between 18 and 65 years | 24 | 0 | 22 | 0 | 19 | 0 | 65
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One family withdrew from IRS control group after random assignment due to displeasure at group assignment and asked for data to be removed.
  years
    number analyzed (Participants) | 24 | 24 | 22 | 22 | 18 | 18 | 128
    (all) | 35.75 (7.56) | 3.80 (1.55) | 35.32 (4.04) | 3.99 (1.55) | 34.56 (6.05) | 4.01 (1.55) | 19.60 (3.74)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One family withdrew from the study after group assignment to IRS Control condition due to dissatisfaction with group assignment and requested all data to be withdrawn.
  Participants
    number analyzed (Participants) | 24 | 24 | 22 | 22 | 18 | 18 | 128
    Female | 20 | 9 | 17 | 5 | 17 | 1 | 69
    Male | 4 | 15 | 5 | 17 | 1 | 17 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: One family withdrew from the study after group assignment to IRS Control condition due to dissatisfaction with group assignment and requested all data to be withdrawn.
  Participants
    Minoritized Race or Ethnicity: number analyzed (Participants) | 24 | 24 | 22 | 22 | 18 | 18 | 128
    Minoritized Race or Ethnicity | 7 | 7 | 5 | 10 | 4 | 5 | 38
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 22 | 22 | 19 | 19 | 130

OUTCOME MEASURES:

1. Primary Outcome: Project ImPACT Intervention Fidelity Checklist
Description: Parents' use of the intervention strategies with their child is measured during a parent-child interaction in the home using the Project ImPACT Intervention Fidelity Checklist (Ingersoll & Dvortcsak, 2019). Parents are asked to (1) play with their child for 10 minutes with a standard set of toys; and (2) have a small snack or meal with their child for 10 minutes. Parents are instructed to interact with their child as they typically would during both activities. Coders rated the parents' use of each of the five Project ImPACT intervention strategies on a scale of 1 ("does not implement the strategy, or almost all attempts to use the strategy are incorrect.") to 5 ("implements the strategy effectively throughout the session"). Scores for each strategy were averaged to form an overall fidelity rating for each activity. Fidelity ratings for each activity were averaged to form the parent fidelity variable.
Time Frame: Post-treatment (6 months)
Population: Analysis of parent data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Parent: Self-Directed Group | Parent: Therapist-Assisted Group | Parent: Information and Resource Support Control Group
Number analyzed (Participants) | 24 | 22 | 18
score on a scale | 2.95 (.15) | 3.62 (.16) | 2.83 (.18)
Statistical Analysis 1: Comparison: Parent: Self-Directed Group vs Parent: Therapist-Assisted Group vs Parent: Information and Resource Support Control Group; The effect of group assignment was examined using MLM, with a significant time X group interaction indicative of an effect of group assignment. Data from T1, T2, and T3 were both used in same analysis; Test type: Superiority; p < .001, Mixed Models Analysis

2. Primary Outcome: Project ImPACT Intervention Fidelity Checklist
Description: as for outcome 1
Time Frame: Follow up (9 months)
Population: Analysis of parent data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Parent: Self-Directed Group | Parent: Therapist-Assisted Group | Parent: Information and Resource Support Control Group
Number analyzed (Participants) | 24 | 22 | 18
score on a scale | 3.12 (.16) | 3.81 (.16) | 2.89 (.19)
Statistical Analysis 1: Comparison: Parent: Self-Directed Group vs Parent: Therapist-Assisted Group vs Parent: Information and Resource Support Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .001, Mixed Models Analysis

3. Primary Outcome: Parent Sense of Competence (PSOC)
Description: The PSOC measures the extent to which parents believe they have the skills and knowledge needed to be good parents (efficacy) and their perceptions regarding the value of parenthood (satisfaction). Parents rated 17 items from 1 ("Strongly disagree") to 6 ("Strongly agree"). Items are summed, with higher scores indicative of higher parenting self-efficacy. Scores can range from 17 to 102, with higher scores indicative of greater self-efficacy
Time Frame: Post-Treatment (6 months)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Parent: Self-Directed Group | Parent: Therapist-Assisted Group | Parent: Information and Resource Support Control Group
Number analyzed (Participants) | 24 | 22 | 18
score on a scale | 74.06 (2.41) | 74.45 (2.44) | 70.76 (2.91)
Statistical Analysis 1: Comparison: Parent: Self-Directed Group vs Parent: Therapist-Assisted Group vs Parent: Information and Resource Support Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .85, Mixed Models Analysis

4. Primary Outcome: Parent Sense of Competence (PSOC)
Description: The PSOC measures the extent to which parents believe they have the skills and knowledge needed to be good parents (efficacy) and their perceptions regarding the value of parenthood (satisfaction). Parents rated 17 items from 1 ("Strongly disagree") to 6 ("Strongly agree"). Items are summed, scores can range from 17 to 102, with higher scores indicative of higher parenting self-efficacy.
Time Frame: Follow up (9 months)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Parent: Self-Directed Group | Parent: Therapist-Assisted Group | Parent: Information and Resource Support Control Group
Number analyzed (Participants) | 24 | 22 | 18
score on a scale | 72.13 (2.37) | 73.15 (2.44) | 69.09 (2.78)
Statistical Analysis 1: Comparison: Parent: Self-Directed Group vs Parent: Therapist-Assisted Group vs Parent: Information and Resource Support Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .85, Mixed Models Analysis

5. Primary Outcome: Weighted Frequency of Intentional Communication
Description: Children's use of intentional communication is scored from a parent-child interaction during play and snack using a modified version of the Weighted Frequency of Intentional Communication (WFIC) coding scheme (Yoder et al., 2021a), which quantifies the maturity of the form and frequency of intentional communication in young children with social communication delays. Coders transcribed and coded all non-imitated communicative utterances, including gestures, contingent vocalizations, single-words, simple phrases, and sentences. Each utterance was weighted (1-4) based on its complexity. Utterances are summed to produce a weighted frequency. Weighted frequency was were converted to a rate per minute by dividing the score by the length of the video. Values were log transformed to improve normality of distribution. Values ranged from -1.30 to 1.57 with higher values indicated higher weighted frequency of intentional communication. Means are adjusted for their T1 measure.
Time Frame: Post-treatment (6 months)
Measure: Mean (Standard Error); unit: log(utterances per minute)
Groups:
- Child: Information and Resource Support Control Group: Child participants will interact with their parent without training in Project ImPACT.
Arm/Group | Child: Self-Directed Group | Child: Therapist-Assisted Group | Child: Information and Resource Support Control Group
Number analyzed (Participants) | 24 | 22 | 18
log(utterances per minute) | .62 (.07) | .64 (.07) | .64 (.08)
Statistical Analysis 1: Comparison: Child: Self-Directed Group vs Child: Therapist-Assisted Group vs Child: Information and Resource Support Control Group; Test type: Superiority; p = .98, ANCOVA

6. Primary Outcome: Child Expressive Language Ability
Description: Equally weighted composite score of child expressive language ability derived from MacArthur Bates Communicative Development Inventory (MB-CDI), Mullen Scales of Early Learning (MSEL) Expressive Language raw score, and Vineland Adaptive Behavior Scales (VABS) Expressive Language raw score. Measures were z-score transformed and averaged. Z-score of 0 represents mean for the participants. Positive z-score represent a better outcome.
Time Frame: Follow up (9 months)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Child: Self-Directed Group | Child: Therapist-Assisted Group | Child: Information and Resource Support Control Group
Number analyzed (Participants) | 24 | 22 | 18
units on a scale | .08 (.12) | -.05 (.12) | -.04 (.13)
Statistical Analysis 1: Comparison: Child: Self-Directed Group vs Child: Therapist-Assisted Group vs Child: Information and Resource Support Control Group; Test type: Superiority; p = .69, ANCOVA

7. Secondary Outcome: Family Impact Questionnaire
Description: Parents complete the 8-item Positive Impact subscale of the Family Impact Questionnaire (FIQ; Donenberg & Baker, 1993) as a measure of their perception of their child's positive impact on their experience as a parent. Parents endorsed items comparing their experience with their child to parents with same-aged typically-developing peers on a 4-point scale; higher sum scores indicate greater positive impact. Scores could range from 8 to 32.
Time Frame: Post-Treatment (6 months)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Parent: Self-Directed Group | Parent: Therapist-Assisted Group | Parent: Information and Resource Support Control Group
Number analyzed (Participants) | 24 | 22 | 18
units on a scale | 22 (1.34) | 23.08 (1.16) | 20.18 (1.36)
Statistical Analysis 1: Comparison: Parent: Self-Directed Group vs Parent: Therapist-Assisted Group vs Parent: Information and Resource Support Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .038, Mixed Models Analysis

8. Secondary Outcome: Parenting Stress Index-Short Form
Description: Parents complete the Parenting Stress Index, Short Form (PSI-SF; Abidin, 1995), a 36-item measure of parenting stress. Parents rated items on a 5-point scale. Items are summed with higher scores indicating greater parenting stress. The Total Stress scale was used as a measure of parenting stress. Raw Scores could range from 36 to 180.
Time Frame: Post-Treatment (6 months)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Parent: Self-Directed Group | Parent: Therapist-Assisted Group | Parent: Information and Resource Support Control Group
Number analyzed (Participants) | 24 | 22 | 18
score on a scale | 92.69 (4.33) | 90.76 (4.39) | 97.50 (5.20)
Statistical Analysis 1: Comparison: Parent: Self-Directed Group vs Parent: Therapist-Assisted Group vs Parent: Information and Resource Support Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .45, Mixed Models Analysis

9. Secondary Outcome: Mullen Scales of Early Learning
Description: The Mullen Scales of Early Learning (MSEL; Mullen, 1995) is a standardized developmental test for young children that assesses skills in expressive language, receptive language, visual reception, and fine motor. The raw score for the Expressive Language scale was used in analyses. Raw scores ranged from 7 to 47. Higher scores indicate better language outcomes. Means are adjusted for their T1 measure.
Time Frame: Follow up (9 months)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Self-Directed Group | Therapist-Assisted Group | Web-Based Information Control Group
Number analyzed (Participants) | 24 | 22 | 18
score on a scale | 23.88 (1.40) | 22.71 (1.90) | 23.12 (1.46)
Statistical Analysis 1: Comparison: Self-Directed Group vs Therapist-Assisted Group vs Web-Based Information Control Group; ANCOVA controlling for T1 measure; Test type: Superiority; p = .92, ANCOVA

10. Secondary Outcome: MacArthur-Bates Communicative Development Inventory
Description: MacArthur-Bates Communicative Development Inventory (MCDI; Fenson et al., 2006) is a parent report instrument that measures early language development, including productive vocabulary. Parents complete either the Words and Gestures Form or Words and Sentences Form, depending on their child's predominant method of communication online. The total number of words parents reported that their child "understands and says" (Words and Gestures Form) or "words produced" (Words and Sentences Form) is used in analyses. Means are adjusted for their T1 measures
Time Frame: Follow up (9 Months)
Measure: Mean (Standard Error); unit: number of words
Arm/Group | Self-Directed Group | Therapist-Assisted Group | Web-Based Information Control Group
Number analyzed (Participants) | 24 | 22 | 18
number of words | 328.68 (31.38) | 270.52 (33.21) | 282.85 (36.73)
Statistical Analysis 1: Comparison: Self-Directed Group vs Therapist-Assisted Group vs Web-Based Information Control Group; ANCOVA controlling for T1 measure; Test type: Superiority; p = .42, ANCOVA

11. Secondary Outcome: Vineland Adaptive Behavior Scales, 2nd Edition
Description: The VABS is a standardized parent interview that assesses adaptive functioning in four domains: communication, socialization, daily living skills, and motor skills. The raw score for the Expressive Language subdomain was used in analyses. Raw scores ranged from 10 to 99. Higher scores indicate better language outcomes. Means are adjusted for their T1 measures
Time Frame: Follow up (9 Months)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Self-Directed Group | Therapist-Assisted Group | Web-Based Information Control Group
Number analyzed (Participants) | 24 | 22 | 18
score on a scale | 48.04 (2.61) | 46.39 (2.72) | 44.30 (3.01)
Statistical Analysis 1: Comparison: Self-Directed Group vs Therapist-Assisted Group vs Web-Based Information Control Group; ANCOVA controlling for T1 measure; Test type: Superiority; p = .65, ANCOVA

12. Other Pre Specified Outcome: Program Engagement
Description: ImPACT Online electronic tracking system. % of learning activities accessed
Time Frame: Post-treatment (6 months)
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Self-Directed Group | Therapist-Assisted Group
Number analyzed (Participants) | 24 | 22
percent | 58.57 (36.93) | 96.29 (7.29)
Statistical Analysis 1: Comparison: Self-Directed Group vs Therapist-Assisted Group; Independent samples t-test; Test type: Superiority; p = .001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Parent: Self-Directed Group | Parent: Therapist-Assisted Group | Parent: Information and Resource Support Control Group | Child: Self-Directed Group | Child: Therapist-Assisted Group | Child: Information and Resource Support Control Group
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/22 | 0/19 | 0/24 | 0/22 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/22 | 0/19 | 0/24 | 0/22 | 0/19
Other Adverse Events (participants affected / at risk) | 0/24 | 0/22 | 0/19 | 0/24 | 0/22 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/81/NCT02721381/Prot_SAP_000.pdf